CLINICAL TRIAL: NCT03248284
Title: Stereological Quantification of Immune-Competent Cells in Biopsies From Painful Achilles Tendons of Psoriatic Arthritis Patients With Ultrasonic Verified Enthesitis: An Exploratory Prospective Cohort Study
Brief Title: Immune-Competent Cell Manifestations in Psoriatic Arthritis Achilles Tendons
Acronym: IMPAACT
Status: Recruiting | Type: Observational
Sponsor: Odense University Hospital (Other)
Collaborators: University of Southern Denmark (Other); Odense Patient Data Explorative Network (Other); The Danish Rheumatism Association (Other); The Psoriasis Association, Denmark (Unknown)
Responsible Party: Principal Investigator, Torkell Ellingsen, Prof MD PhD, Odense University Hospital
Other Study IDs: OUH-IMPAACT-02
Record Dates: First submitted 2017-08-09; First posted 2017-08-14 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-03

CONDITIONS: Psoriatic Arthritis; Enthesitis
MeSH Terms: conditions — Arthritis, Psoriatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Achilles tendon tissue specimens, blood- and fecal samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Tendon biopsy procedure — Two tendon biopsy specimens will be obtained from one Achilles tendon with enthesitis.

SUMMARY:
Tendon pathologies (enthesitis) are a characteristic component of psoriatic arthritis (PsA), and are observed in 35% to 50% of PsA patients. The Achilles tendon is one of the most commonly affected sites. This condition often causes great morbidity and loss of quality of life, and response only suboptimal to current intervention strategies. One of the main obstacles for the development of effective treatment methods is that the disease mechanisms remain poorly understood. To our knowledge, no one has yet ascertained the presence and function of immune-competent cells and inflammatory markers in tendons tissue from PsA patients suffering from Achilles enthesitis.

DETAILED DESCRIPTION:
Aim: The main objective of the IMPAACT study is to describe the histological findings of PsA Achilles enthesitis, and to a) Characterize and b) Quantify the immune-competent cell presence in tendon specimens obtained from the mid-portion and entheseal site of the Achilles tendon from PsA patients with enthesitis using immunohistochemistry and a stereological technique for the quantification. And secondly, to compare these observations with a) Those in healthy Achilles tendons, and b) Those in mono-symptomatic, non-PsA, chronic Achilles tendinopathy. Secondly, to examine whether one or more of the immune-competent cell types in the PsA tendons are associated with 3-months remission rate of Achilles tendon pain, or with baseline a) Ultrasonic findings of the Achilles tendon; b) PsA disease activity; c) Tendon protein analyses; d) Risk factors of cardiovascular disease; e) Blood biomarkers of systemic inflammation; and f) Fecal microbiota composition.

Methods: This study (IMPAACT) is a prospective, cohort study including 30 PsA patients (fulfilling the the Classification Criteria for Psoriatic Arthritis (CASPAR criteria)) with pain at the Achilles tendon insertion. At baseline, all participants will be examined clinically regarding overall PsA disease activity (Psoriasis Area Severity Index (PASI skin score), the Research Consortium of Canada (SPARCC) Enthesitis score, swollen/tender joint count) and asked to fill out a questionnaire consisting of the validated Scandinavian (Danish) version of the Victorian Institute of Sport Assessment of Achilles tendons (VISA-A) in addition to a study-composed questionnaire comprising general questions regarding patient characteristics. An ultrasonic examination of the Achilles tendons will be performed before ultrasound guided Achilles tendon specimens will be obtained from the most painful Achilles tendon. Tendon samples will be evaluated immunohistochemically by quantifying the presence of macrophages (CD68-KP1+), T-lymphocytes (CD3+), B-lymphocytes (CD20+), natural killer cells (CD56+), neutrophils (granzyme-B+), mast cells and inflammatory markers using a stereological technique. Also, a protein analysis of the tendon tissue will be conducted. Venous blood will be analysed for levels of systemic inflammatory markers, as well as screened for cardiovascular risk factors including dyslipidaemia, and diabetes. After the baseline examination, all participants will be treated and monitored in accordance with the Danish national guideline recommendations for PsA patients. A 3-months follow-up examination will be performed to determine the remission status of the Achilles tendon pain. Data will be analysed using the STATA statistical package.

Conclusion: PsA is a painful and debilitating inflammatory disease. The current treatment remains suboptimal. We hope to provide new insight into the cellular mechanisms underlying PsA tendon and enthesis pathologies.

ELIGIBILITY:
Inclusion Criteria:

* Fulfilling the CASPAR criteria
* Insertional Achilles tendon pain
* Ultrasonic findings of inflammatory disease at the painful Achilles tendon insertion (= enthesitis) defined as abnormally hypoechoic (loss of normal fibrillar architecture) and/or thickened tendon at its bony attachment, seen in two perpendicular planes that may exhibit a Doppler signal or bony changes, including enthesophytes, and erosions.

Exclusion Criteria:

* Other inflammatory rheumatic diseases than PsA
* Ultrasonic signs of complete rupture of the Achilles tendon
* Not wishing to participate or not suited for project evaluation

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Psoriatic arthritis patients with Achilles enthesitis.
  There will be no restrictions regarding previous or current local and/or systemic anti-inflammatory treatments, however, any type of such treatment will be registered and used to stratify patients into treatment groups for the statistical analysis. Patients who have never received any systemic and/or local anti-inflammatory treatment will be referred to as treatment naïve.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2017-08-21 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Presence of Immune-competent cells and inflammatory markers | Baseline
  CD3, CD4, CD8, CD20, CD34 (or CD31), CD56, S100 beta (CD57), CD68 (PGM1) or CD163, TNF-alfa, IL-6, IL-23 and other inflammatory markers.

SECONDARY OUTCOMES:
Protein analyses | Baseline
  Protein analyses performed on Achilles tendon tissue
Adverse events | From baseline to 3-month follow-up
  Number of adverse events during follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Maja S Kragsnaes, MD PhDfellow, Principal Investigator — Odense University Hospital
Locations (2):
- Denmark (2):
  - Odense University Hospital, Odense
  - Diagnostic Center, Silkeborg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McGonagle DG, Helliwell P, Veale D. Enthesitis in psoriatic disease. Dermatology. 2012;225(2):100-9. doi: 10.1159/000341536. Epub 2012 Oct 27. PMID 23108016
- [Background] Terslev L, Naredo E, Iagnocco A, Balint PV, Wakefield RJ, Aegerter P, Aydin SZ, Bachta A, Hammer HB, Bruyn GA, Filippucci E, Gandjbakhch F, Mandl P, Pineda C, Schmidt WA, D'Agostino MA; Outcome Measures in Rheumatology Ultrasound Task Force. Defining enthesitis in spondyloarthritis by ultrasound: results of a Delphi process and of a reliability reading exercise. Arthritis Care Res (Hoboken). 2014 May;66(5):741-8. doi: 10.1002/acr.22191. PMID 24151222
- [Background] Khan KM, Cook JL, Bonar F, Harcourt P, Astrom M. Histopathology of common tendinopathies. Update and implications for clinical management. Sports Med. 1999 Jun;27(6):393-408. doi: 10.2165/00007256-199927060-00004. PMID 10418074
- [Background] Fredberg U, Stengaard-Pedersen K. Chronic tendinopathy tissue pathology, pain mechanisms, and etiology with a special focus on inflammation. Scand J Med Sci Sports. 2008 Feb;18(1):3-15. doi: 10.1111/j.1600-0838.2007.00746.x. PMID 18294189
- [Background] Ryan C, Korman NJ, Gelfand JM, Lim HW, Elmets CA, Feldman SR, Gottlieb AB, Koo JY, Lebwohl M, Leonardi CL, Van Voorhees AS, Bhushan R, Menter A. Research gaps in psoriasis: opportunities for future studies. J Am Acad Dermatol. 2014 Jan;70(1):146-67. doi: 10.1016/j.jaad.2013.08.042. Epub 2013 Oct 11. PMID 24126079
- [Background] Jacques P, Lambrecht S, Verheugen E, Pauwels E, Kollias G, Armaka M, Verhoye M, Van der Linden A, Achten R, Lories RJ, Elewaut D. Proof of concept: enthesitis and new bone formation in spondyloarthritis are driven by mechanical strain and stromal cells. Ann Rheum Dis. 2014 Feb;73(2):437-45. doi: 10.1136/annrheumdis-2013-203643. Epub 2013 Aug 6. PMID 23921997
- [Background] Kragsnaes MS, Fredberg U, Stribolt K, Kjaer SG, Bendix K, Ellingsen T. Stereological quantification of immune-competent cells in baseline biopsy specimens from achilles tendons: results from patients with chronic tendinopathy followed for more than 4 years. Am J Sports Med. 2014 Oct;42(10):2435-45. doi: 10.1177/0363546514542329. Epub 2014 Jul 31. PMID 25081311
- [Background] McGonagle D, Marzo-Ortega H, O'Connor P, Gibbon W, Hawkey P, Henshaw K, Emery P. Histological assessment of the early enthesitis lesion in spondyloarthropathy. Ann Rheum Dis. 2002 Jun;61(6):534-7. doi: 10.1136/ard.61.6.534. PMID 12006328